CLINICAL TRIAL: NCT07040839
Title: Comparative Efficacy of Omeprazole and Vonoprazan in the Treatment of Helicobacter Pylori Infection
Brief Title: Comparison of Omeprazole vs Vonoprazon in Treatment of H Pylori Infection
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Wajeeha Qayyum, Consultant/Assistant Professor Medicine, Rehman Medical Institute - RMI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMI/RMI-REC/approval 182
Record Dates: First submitted 2025-06-12; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: H Pylori
Keywords: omeprazole; vonoprazon; proton pump inhibitors
MeSH Terms: interventions — Clarithromycin; Amoxicillin; Omeprazole; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- First-Line Therapy with Omeprazole (Experimental)
  Interventions: Drug: Clarithromycin 500 mg; Drug: Amoxicillin 1 g; Drug: Omeprazole 40 mg
- First-Line Therapy with Vonoprazan (Experimental)
  Interventions: Drug: Clarithromycin 500 mg; Drug: Amoxicillin 1 g; Drug: Vonoprazan 20 mg
- Second-Line Therapy with Omeprazole (Experimental)
  Interventions: Drug: Levofloxacin 500 mg; Drug: Amoxicillin 1 g; Drug: Omeprazole 40 mg
- Second-Line Therapy with Vonoprazan (Experimental): Participants receiving second-line therapy (levofloxacin + amoxicillin) with vonoprazan as the acid suppressant.
  Interventions: Drug: Levofloxacin 500 mg; Drug: Amoxicillin 1 g; Drug: Vonoprazan 20 mg

INTERVENTIONS:
Drug: Clarithromycin 500 mg — Clarithromycin 500 mg orally twice daily for 14 days
  Arms: First-Line Therapy with Omeprazole
Drug: Amoxicillin 1 g — Omeprazole 40 mg orally twice daily for 14 days, then 40 mg once daily for 4 weeks
  Arms: First-Line Therapy with Omeprazole
Drug: Omeprazole 40 mg — Omeprazole 40 mg orally twice daily for 14 days, then 40 mg once daily for 4 weeks
  Arms: First-Line Therapy with Omeprazole
Drug: Clarithromycin 500 mg — Clarithromycin 500 mg orally twice daily for 14 days
  Arms: First-Line Therapy with Vonoprazan
Drug: Amoxicillin 1 g — Amoxicillin 1 g orally twice daily for 14 days
  Arms: First-Line Therapy with Vonoprazan
Drug: Vonoprazan 20 mg — Vonoprazan 20 mg orally twice daily for 14 days, then 20 mg once daily for 4 weeks
  Arms: First-Line Therapy with Vonoprazan
Drug: Levofloxacin 500 mg — Levofloxacin 500 mg orally once daily for 14 days
  Arms: Second-Line Therapy with Omeprazole
Drug: Amoxicillin 1 g — Amoxicillin 1 g orally twice daily for 14 days
  Arms: Second-Line Therapy with Omeprazole
Drug: Omeprazole 40 mg — Omeprazole 40 mg orally twice daily for 14 days, then 40 mg once daily for 4 weeks
  Arms: Second-Line Therapy with Omeprazole
Drug: Levofloxacin 500 mg — Levofloxacin 500 mg orally once daily for 14 days
  Arms: Second-Line Therapy with Vonoprazan
Drug: Amoxicillin 1 g — Amoxicillin 1 g orally twice daily for 14 days
  Arms: Second-Line Therapy with Vonoprazan
Drug: Vonoprazan 20 mg — Vonoprazan 20 mg orally twice daily for 14 days, then 20 mg once daily for 4 weeks
  Arms: Second-Line Therapy with Vonoprazan

SUMMARY:
Current studies have primarily focused on comparing the advantages and disadvantages of P-CAB and PPI drugs, with little comparison between different P-CAB drugs or between regimens with varying drug combinations and treatment durations.

This study aims to evaluate the clinical effectiveness of vonoprazan-based H. pylori eradication therapy and compare it to that of conventional PPI based therapy in clinical practice.

DETAILED DESCRIPTION:
Currently, there are numerous H. pylori eradication regimens, but opinions vary regarding the effectiveness of those based on P-CAB or PPI. Zhang et al. 4 concluded that the P-CAB-based triple regimen was superior to the PPI-based regimen, whereas Du et al.5 suggested that a vonoprazan and amoxicillin duo regimen may be the preferred first-line option for H. pylori eradication in clinical practice. However, due to limited evidence, the efficacy of various H. pylori eradication regimens using tegoprazan or vonoprazan could not be compared.

Current studies have primarily focused on comparing the advantages and disadvantages of P-CAB and PPI drugs, with little comparison between different P-CAB drugs or between regimens with varying drug combinations and treatment durations.

This study aims to evaluate the clinical effectiveness of vonoprazan-based H. pylori eradication therapy and compare it to that of conventional PPI based therapy in clinical practice.

Objective: To compare the efficacy of vonoprazan-based H. pylori eradication therapy with conventional proton pump inhibitors based therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who tested positive on stool antigen

Exclusion Criteria:

* patients under 12 years old.
* Patients who have penicillin allergy.
* Patients who have underlying dysrhythmia forbidding the use of macrolide -. Patient who have hypersensitivity to any of these antibiotics or proton pump inhibitors.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
H. pylori Eradication Rate | 4-6 weeks after completion of therapy
  Proportion of participants with successful eradication of Helicobacter pylori infection, confirmed by a negative stool antigen test.

SECONDARY OUTCOMES:
Incidence of Adverse Events | During the 6-week treatment and follow-up period
  Number and type of treatment-related adverse effects (e.g., nausea, diarrhea, headache, abdominal discomfort) reported by participants during or after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Rehman Medical Institue, Peshawar, K, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Malfertheiner P, Moss SF, Daniele P, Pelletier C, Jacob R, Tremblay G, Hubscher E, Leifke E, Chey WD. Potassium-Competitive Acid Blocker and Proton Pump Inhibitor-Based Regimens for First-Line Helicobacter pylori Eradication: A Network Meta-Analysis. Gastro Hep Adv. 2022 Jun 17;1(5):824-834. doi: 10.1016/j.gastha.2022.06.009. eCollection 2022. PMID 39131848
- [Background] Du RC, Hu YX, Ouyang Y, Ling LX, Xu JY, Sa R, Liu XS, Hong JB, Zhu Y, Lu NH, Hu Y. Vonoprazan and amoxicillin dual therapy as the first-line treatment of Helicobacter pylori infection: A systematic review and meta-analysis. Helicobacter. 2024 Jan-Feb;29(1):e13039. doi: 10.1111/hel.13039. Epub 2023 Nov 30. PMID 38036941
- [Background] Zhang M, Pang M, Zhang M. Efficacy and safety of potassium-competitive acid blockers versus proton pump inhibitors as Helicobacter pylori eradication therapy: a meta-analysis of randomized clinical trials. Clinics (Sao Paulo). 2022 Jul 7;77:100058. doi: 10.1016/j.clinsp.2022.100058. eCollection 2022. PMID 35810638
- [Background] Kim GH. Proton Pump Inhibitor-Related Gastric Mucosal Changes. Gut Liver. 2021 Sep 15;15(5):646-652. doi: 10.5009/gnl20036. PMID 32327613
- [Background] Kiyotoki S, Nishikawa J, Sakaida I. Efficacy of Vonoprazan for Helicobacter pylori Eradication. Intern Med. 2020 Jan 15;59(2):153-161. doi: 10.2169/internalmedicine.2521-18. Epub 2019 Jun 27. PMID 31243237
- [Background] Sun Y, Zhang J. Helicobacter pylori recrudescence and its influencing factors. J Cell Mol Med. 2019 Dec;23(12):7919-7925. doi: 10.1111/jcmm.14682. Epub 2019 Sep 19. PMID 31536675